CLINICAL TRIAL: NCT01184339
Title: Prospective Study Into the Performance of the MicroPhage S. Aureus/MSSA/MRSA Test Direct From Blood Culture Positives
Status: Completed | Type: Observational
Sponsor: MicroPhage, Inc. (Industry)
Responsible Party: Drew Smith, Ph.D., MicroPhage, Inc.
Other Study IDs: MP2009-B
Record Dates: First submitted 2010-03-04; First posted 2010-08-18 (Estimated); Last update posted 2010-08-18 (Estimated); Status verified 2010-08

CONDITIONS: Bacteremia
Keywords: Staphylococcus; aureus; methicillin; resistant; MRSA; MSSA; Blood Culture; diagnostic
MeSH Terms: conditions — Bacteremia; Disease

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Approximately 100 uL of deidentified blood culture sample per test sample run.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Standard of Care: Current practice methods for the determination of bacteremia, specific to site practice.
  Interventions: Device: MicroPhage S. aureus/MSSA/MRSA Blood Culture Test
- Gold Standard ID/AST: Identification of S. aureus: coagulase positive, catalase positive, Staphaurex positive, and PYR negative, if performed).
  Determination of MRSA:S. aureus gold standard and </=11mm OXA DD or </=21mm CFX DD.
  Determination of MSSA: S. aureus gold standard and >/=13mm OXA DD or >/=22mm CFX DD.
  Interventions: Device: MicroPhage S. aureus/MSSA/MRSA Blood Culture Test

INTERVENTIONS:
Device: MicroPhage S. aureus/MSSA/MRSA Blood Culture Test — In vitro diagnostic for the Identification of S. aureus and determination of MSSA or MRSA from a positive blood culture.
  Approximately 5 hour rapid test.

SUMMARY:
Direct in-vitro identification of S. aureus, methicillin-sensitive S. aureus (MSSA), and methicillin-resistant S. aureus (MRSA) from positive blood cultures by MicroPhage's bacteriophage-based diagnostic platform, two gold-standard reference methods, and two predicate devices with similar indications for use.

DETAILED DESCRIPTION:
This is a multi-center, FDA clinical study designed to investigate the safety and performance of the MicroPhage S. aureus/MSSA/MRSA test direct from blood culture positives. Informed consent is not anticipated, as this is a laboratory performance study with no patient intervention. The MicroPhage Test will be compared to site standards of care, market-available rapid tests, two predicate tests, and two disk diffusion tests for antimicrobial susceptibility. The study will last approximately 4-6 months (Bactec), dependent on the accrual rate of each institution.

This study is designed to support the following product indications for use:

The MicroPhage S. aureus/MSSA/MRSA Blood Culture Test is a qualitative in vitro diagnostic test for the rapid identification of Staphylococcus aureus and determination of methicillin susceptibility (MSSA) or methicillin resistance (MRSA) directly from positive blood cultures.

The test uses bacteriophage amplification to rapidly and phenotypically identify the presence of S. aureus and assess the response of the target organism to cefoxitin as an analog to methicillin.

This test is performed on positive blood cultures.

Subculturing of positive blood cultures is necessary for further susceptibility test determinations.

Results of the study analysis will be in the form of descriptive statistics (mean, median, standard deviation, frequencies) for all study variables. Associations among variables will be presented using correlation coefficients, as well as odds ratios and parameter estimates from multivariable regression (linear and logistic) where applicable.

ELIGIBILITY:
Inclusion Criteria:

* Blood culture positive samples from subjects aged 18+, with any of the following bottle types:
* BD Bactec Standard Aerobic and Anaerobic,
* BD Bactec Plus Aerobic and Anaerobic,
* Completion of the MicroPhage test protocol on the sample.

Exclusion Criteria:

* Samples from subjects under 18 years of age,
* Samples from any other not included bottle types,
* Samples from blood culture positives over 24 hours from alarm,
* Samples deemed contaminated,
* Mislabeled / misidentified samples or data without documented corrections,
* Violations and/or deviations from the MicroPhage test protocol and/or other included test protocols under study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital patients with at least one positive blood culture.
Sampling Method: Non-Probability Sample
Enrollment: 1165 (Actual)
Dates: Start 2009-08; Primary Completion 2010-01 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Determination of the performance of the MicroPhage S. aureus/ MSSA/MRSA Test for identification of S. aureus and determination of MRSA and MSSA direct from clinical blood culture positives against gold standard laboratory tests. | Daily per device protocol
  i) Comparison of the MicroPhage S. aureus/MSSA/MRSA test for identification of S. aureus to the gold Standard for S. aureus (coagulase positive, catalase positive, Staphaurex positive, and PYR negative).
Determination of comparative performance of the MicroPhage S. aureus/MRSA/MSSA Test to the Oxoid PBP2a for determination of MRSA. | Daily per device protocol
  Performance comparison of the two tests.
Determination of the performance of the MicroPhage S. aureus/ MSSA/MRSA Test for identification of S. aureus and determination of MRSA and MSSA direct from clinical blood culture positives against gold standard laboratory tests. | Daily per device protocol
  ii) Comparison of the MicroPhage S. aureus/MSSA/MRSA test for identification of S. aureus and determination of MRSA to the gold Standard for MRSA (S. aureus gold standard and </=10mm OXA DD or </=21mm CFX DD) iii) Comparison of the MicroPhage S. aureus/MSSA/MRSA test for identification of S. aureus and determination of MSSA to the gold Standard for MSSA (S. aureus gold standard and >/=13mm OXA DD or >/=22mm CFX DD)

SECONDARY OUTCOMES:
Determination of clinical performance of the MicroPhage S. aureus/MSSA/MRSA Test to monitor S. aureus/MSSA/MRSA bacteremia clinical blood culture positives with unique subjects. | Daily per device protocol
  Study of MicroPhage Test performance to primary endpoint criteria with one sample per unique subject.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kirn, MD.PhD, Principal Investigator — Rutgers, The State University of New Jersey; Chao Qi, PhD, Principal Investigator — Northwestern Medical School; Barth Reller, MD, Principal Investigator — Duke Medical College; Connie Savor-Price, MD, Principal Investigator — Denver Health